CLINICAL TRIAL: NCT00023166
Title: Phase I Study of PEG-Paclitaxel In Patients With Advanced Solid Tumors and Lymphomas
Brief Title: Phase I Study of PEG-Paclitaxel In Patients With Advanced Solid Tumors & Lymphomas
Status: Terminated | Phase: Phase 1 | Type: Interventional
Sponsor: Enzon Pharmaceuticals, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTX-5001
Record Dates: First submitted 2001-08-24; First posted 2001-08-27 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2004-03

CONDITIONS: Neoplasm; Lymphomas; Neoplasm Metastasis
Keywords: Phase I; Open label; Safety/efficacy; Lymphomas; Advanced primary and/or metastatic solid tumors; Neoplasms; Neoplasm metastasis
MeSH Terms: conditions — Neoplasms; Lymphoma; Neoplasm Metastasis | interventions — poly(ethylene glycol)-conjugated paclitaxel-2'-glycinate

INTERVENTIONS:
Drug: PEG-paclitaxel

SUMMARY:
Studies of PEG-paclitaxel have been terminated

ELIGIBILITY:
None - Study has been terminated.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-05; Study Completion 2002-05